CLINICAL TRIAL: NCT00460655
Title: A Multicenter Study to Evaluate the Efficacy and Safety in Patients With Post-Stroke Lower Limb Spasticity Receiving a Double-Blind, Placebo-Controlled GSK1358820 Treatment Followed by an Open-Label GSK1358820 Treatment
Brief Title: Study of GSK1358820 In Patients With Post-Stroke Lower Limb Spasticity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTX108512
Record Dates: First submitted 2007-04-13; First posted 2007-04-16 (Estimated); Results first posted 2010-01-26 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-08

CONDITIONS: Post-Stroke Spasticity; Cerebrovascular Accident
Keywords: Post-Stroke; Lower Limb; botulinum toxin type A; Spasticity
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BTX (Active Comparator)
  Interventions: Drug: GSK1358820
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK1358820 — botulinum toxin type A
  Arms: BTX
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a study to confirm the superior efficacy of GSK1358820 over placebo in patients with equinus deformity associated with post-stroke lower limb spasticity using the Modified Ashworth Scale (MAS) ankle score.

DETAILED DESCRIPTION:
This is a study to confirm the superior efficacy of GSK1358820 over placebo in patients with equinus deformity associated with post-stroke lower limb spasticity using the Modified Ashworth Scale (MAS) ankle score.

ELIGIBILITY:
Inclusion Criteria:

* Subjects eligible for enrollment in the study must meet all of the following criteria:
* Patients with lower limb spasticity who are at least 6 months post-stroke and present with equinus deformity (plantar flexion of the ankle) at the start of double-blind phase (Visit 2).
* Patients with MAS ankle score of ≥3 at the start of double-blind phase (Visit 2).
* Male or female between 20 and 80 years of age at the time of informed consent. For males, only those who can practice contraception during the study period are eligible.
* ≥50kg in weight at the start of double-blind phase (Visit 2).
* Inpatient or outpatient; however, the hospitalization status must remain unchanged during the double-blind phase. NOTE: Subjects may be hospitalized for ≤10 days after injection during the treatment period.
* Written informed consent from the subject him/herself. If the subject's signature is not legible, the attendance of a witness is required.

Exclusion Criteria:

* A subject will not be eligible for inclusion in this study if any of the following criteria apply:
* Bilateral hemiplegia or quadriplegia.
* Presence of fixed contractures of the ankle (absence of range of motion).
* Profound atrophy of the muscles to be injected.
* Previous surgical intervention, phenol block, ethanol block, or Muscle Afferent Block (MAB) for ankle spasticity.
* Casting of the study lower limb within 3 months prior to the start of double-blind phase (Visit 2).
* Current treatment with intrathecal baclofen.
* Use of peripheral muscle relaxants (dantrolene sodium, suxamethonium chloride, pancuronium bromide, vecuronium bromide, rocuronium bromide).
* Concurrent use of antibiotics that interfere with neuromuscular transmission, such as aminoglycoside antibiotics (e.g., streptomycin sulfate, kanamycin sulfate, gentamicin sulfate, neomycin sulphate, spectinomycin hydrochloride), polypeptide antibiotics (e.g., polymixin B sulfate), lincomycin antibiotics (e.g., lincomycin hydrochloride, clindamycin), and enviomycin sulfate.
* Previous or current botulinum toxin therapy of any serotype.
* Diagnosis of systemic neuromuscular disorders (e.g., myasthenia gravis, Lambert-Eaton syndrome, amyotrophic lateral sclerosis).
* Females who are pregnant, nursing, may be pregnant, or planning a pregnancy during the study period.
* Known allergy or hypersensitivity to any ingredient of study medication (e.g., human serum albumin).
* Presence of psychiatric disorder or impairment of intellectual function that may interfere with the subject's ability to give informed consent or the conduct of the study.
* Bedridden patients.
* Presence of clinically unstable severe cardiovascular disease.
* Presence of clinically significant severe renal or hepatic disease.
* Infection or dermatological condition at the proposed injection sites.
* Previous or planned participation in another clinical study (including the upper limb spasticity study of GSK1358820) within 6 months prior to the start of double-blind phase (Visit 2).
* Others whom the investigator or sub investigator considers not eligible for the study.
* Clinically significant severe reduction of muscle strength.
* Angle closure glaucoma or its preposition (narrow angle).

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- Japan (9):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Yamaguchi

REFERENCES:
- [Derived] Kaji R, Osako Y, Suyama K, Maeda T, Uechi Y, Iwasaki M; GSK1358820 Spasticity Study Group. Botulinum toxin type A in post-stroke lower limb spasticity: a multicenter, double-blind, placebo-controlled trial. J Neurol. 2010 Aug;257(8):1330-7. doi: 10.1007/s00415-010-5526-3. Epub 2010 Apr 1. PMID 20358216

RESULTS

PARTICIPANT FLOW:
Groups:
- BTX 300U: BTX (GSK1358820) 300U (24 mL) was injected into the lower limb muscles in the 12-week double-blind phase (DB) (once at Week 0)
- Placebo: Placebo 24 mL was injected into the lower limb muscles in the 12-week double-blind phase (DB) (once at Week 0)
- DB BTX + OL BTX: BTX (GSK1358820) 300U (24 mL) was injected into the lower limb muscles in the 12-week double-blind phase (DB) (once at Week 0) plus the 36-week open-label phase (OL) following the DB phase (up to 3 times, from Week 12 to Week 36 if participant met re-injection criteria [Modified Ashworth Scale (MAS) score of ankle >=2 and at least 12 weeks (84 days) since the last injection])
- DB Placebo + OL BTX: Placebo 24 mL was injected into the lower limb muscles in the 12-week double-blind phase (DB) (once at Week 0) plus BTX (GSK1358820) 300U in open-label phase (OL) following the DB phase (up to 3 times, from Week 12 to Week 36 if participant met re-injection criteria [Modified Ashworth Scale (MAS) score of ankle >=2 and at least 12 weeks (84 days) since the last injection])
Period: Double-Blind Phase (12 Weeks)
Arm/Group | BTX 300U | Placebo | DB BTX + OL BTX | DB Placebo + OL BTX
Started | 58 | 62 | 0 | 0
Completed | 52 | 61 | 0 | 0
Not Completed | 6 | 1 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Period: Open-Label Phase (36 Weeks)
Arm/Group | BTX 300U | Placebo | DB BTX + OL BTX | DB Placebo + OL BTX
Started | 0 | 0 | 52 | 61
Completed | 0 | 0 | 45 | 52
Not Completed | 0 | 0 | 7 | 9
Not completed — Adverse Event | 0 | 0 | 1 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 6 | 2
Not completed — Meeting the Exclusion Criteria | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BTX 300U | Placebo | Total
Number analyzed (Participants) | 58 | 62 | 120
Age Continuous [Mean (Standard Deviation); unit: years] | 62.4 (8.66) | 62.5 (9.32) | 62.5 (8.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 16 | 24
  Male | 50 | 46 | 96
Race/Ethnicity, Customized [Number; unit: participants]
  Asian-Japanese | 58 | 62 | 120

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve (AUC) for the Change From Baseline in Modified Ashworth Scale (MAS) Ankle Score to the End of the DB Phase (Week 12)
Description: Change from baseline in MAS ankle score using a 6-point scale (0, 1, 1+ [regarded as 1.5], 2, 3, and 4; 0=no increase in muscle tone; 4=affected part[s] rigid in flexion/extension) to each time point in the DB phase was calculated. In the graph plotting time points on the horizontal axis and changes from baseline on the vertical axis, the area surrounded by the MAS ankle score change curve and the horizontal axis was calculated and used as a summary index (AUC) for assessment of the MAS ankle score. Negative changes from baseline indicate improvement, and the AUC has a negative sign.
Time Frame: Baseline, Week 12
Population: Full Analysis Set (FAS): all participants randomized, with the exception of those who did not receive any investigational product and those with no assessment of post-treatment MAS ankle score
Measure: Mean (Standard Deviation); unit: Score*week
Arm/Group | BTX 300U | Placebo
Number analyzed (Participants) | 58 | 62
Score*week | -8.513 (6.6904) | -5.085 (6.6496)
Statistical Analysis 1: Comparison: BTX 300U vs Placebo; Test type: Superiority or Other; p = 0.006, t-test, 2 sided; Mean Difference (Net) = -3.428, 95% CI [-5.841 to -1.016]

2. Secondary Outcome: Mean Change From Baseline in the MAS Ankle Score From Baseline to Week 12 of the Double-blind Phase
Description: The investigator assessed Modified Ashworth Scale (MAS) ankle score using a 6-point scale (0, 1, 1+, 2, 3, and 4; 0=No increase in muscle tone to 4=Affected part[s] rigid in flexion or extension) at each time point in the double-blind phase. The "+1" (slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder [less than half] of ROM [range of motion]) of MAS score is regarded as score 1.5.
Time Frame: Baseline; Weeks 1, 4, 6, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | BTX 300U | Placebo
Number analyzed (Participants) | 58 | 62
Points on a scale
  Week 1 | -0.61 (0.675) | -0.52 (0.765)
  Week 4 | -0.88 (0.687) | -0.43 (0.718)
  Week 6 | -0.91 (0.733) | -0.47 (0.712)
  Week 8 | -0.82 (0.660) | -0.43 (0.676)
  Week 12 | -0.56 (0.685) | -0.40 (0.583)

3. Secondary Outcome: Mean Change From Baseline in the Physician's Rating Score (PRS) From Baseline to Week 12 of the Double-blind Phase
Description: The investigator assessed the PRS of gait pattern consisting of 3 parameters. Affected limb was scored on a scale of -1 (worst) to 9 (best) based on 3 parameters (initial foot contact, foot contact at midstance, gait assistive devices) at each time point in double-blind phase.
Time Frame: Baseline; Weeks 1, 4, 6, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | BTX 300U | Placebo
Number analyzed (Participants) | 58 | 62
Points on a scale
  Week 1 | 0.40 (1.178) | 0.66 (1.401)
  Week 4 | 0.54 (1.224) | 0.63 (1.449)
  Week 6 | 0.46 (1.190) | 0.72 (1.474)
  Week 8 | 0.61 (1.188) | 0.78 (1.811)
  Week 12 | 0.55 (1.264) | 0.58 (1.565)

4. Secondary Outcome: Mean Change From Baseline in the Time (Seconds) to Walk 10 Meters From Baseline to Week 12 of the Double-blind Phase
Description: The time (seconds) required to walk 10 meters was measured at each time point in the double-blind phase.
Time Frame: Baseline; Weeks 1, 4, 6, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | BTX 300U | Placebo
Number analyzed (Participants) | 58 | 62
seconds
  Week 1 | 2.14 (34.828) | -5.02 (11.436)
  Week 4 | -6.10 (22.852) | -7.37 (20.782)
  Week 6 | -7.80 (20.568) | -8.48 (18.075)
  Week 8 | -3.14 (35.780) | -8.19 (18.633)
  Week 12 | -10.14 (26.930) | -8.53 (24.710)

5. Secondary Outcome: Mean Change From Baseline in the Clinical Global Impression (CGI) Score of Functional Disability Assessed by the Investigator From Baseline to Week 12 of the Double-blind Phase
Description: The CGI of functional disability was assessed at each visit using the 11-point Numeric Rating Scale (NRS) (-5=Worst Possible to 5=Best Possible) at each time point in the double-blind phase.
Time Frame: Baseline; Weeks 1, 4, 6, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | BTX 300U | Placebo
Number analyzed (Participants) | 58 | 62
Points on a scale
  Week 1 | 0.82 (1.283) | 0.45 (1.082)
  Week 4 | 1.09 (1.254) | 0.64 (1.065)
  Week 6 | 1.21 (1.558) | 0.66 (1.182)
  Week 8 | 1.13 (1.318) | 0.59 (1.230)
  Week 12 | 0.81 (1.302) | 0.52 (1.273)

6. Secondary Outcome: Mean Change From Baseline in the Clinical Global Impression (CGI) Score of Functional Disability Assessed by the Participant From Baseline to Week 12 of the Double-blind Phase
Description: as for outcome 5
Time Frame: Baseline; Weeks 1, 4, 6, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | BTX 300U | Placebo
Number analyzed (Participants) | 58 | 62
Points on a scale
  Week 1 | 0.49 (1.477) | 0.34 (1.470)
  Week 4 | 0.75 (1.575) | 0.44 (1.756)
  Week 6 | 0.82 (1.850) | 0.72 (1.976)
  Week 8 | 1.00 (2.028) | 0.70 (1.978)
  Week 12 | 0.49 (1.527) | 0.49 (2.180)

7. Secondary Outcome: Mean Change From Baseline in the Clinical Global Impression (CGI) Score of Functional Disability Assessed by the Physiotherapist/Occupational Therapist From Baseline to Week 12 of the Double-blind Phase
Description: as for outcome 5
Time Frame: Baseline; Weeks 1, 4, 6, 8, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | BTX 300U | Placebo
Number analyzed (Participants) | 58 | 62
Points on a scale
  Week 1 | 0.63 (1.190) | 0.48 (1.004)
  Week 4 | 0.64 (1.271) | 1.07 (1.377)
  Week 6 | 0.82 (1.550) | 1.03 (1.906)
  Week 8 | 1.04 (1.780) | 1.00 (1.643)
  Week 12 | 1.02 (1.337) | 0.97 (1.505)

8. Secondary Outcome: Mean Change From Baseline (at the Start of the Double-blind Phase) in the MAS Ankle Score at 4, 8, and 12 Weeks After Each Injection in the Open-label Phase
Description: The investigator assessed Modified Ashworth Scale (MAS) ankle score using a 6-point scale (0, 1, 1+, 2, 3, and 4; 0=No increase in muscle tone to 4=Affected part[s] rigid in flexion or extension) at each time point from baseline (at the start of the double-blind phase) to Week 48. The "+1" (slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder [less than half] of ROM [range of motion]) of MAS score is regarded as score 1.5.
Time Frame: Baseline; Weeks 4, 8, and 12 after each injection (up to Week 48; injections given from Week 12 to Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | DB BTX + OL BTX | DB Placebo + OL BTX
Number analyzed (Participants) | 50 | 57
Points on a scale
  Week 4 after first injection in OL | -1.37 (0.660) | -1.27 (0.653)
  Week 8 after first injection in OL | -1.29 (0.682) | -1.33 (0.590)
  Week 12 after first injection in OL | -1.03 (0.646) | -1.04 (0.654)
  Week 4 after second injection in OL | -1.55 (0.706) | -1.51 (0.640)
  Week 8 after second injection in OL | -1.36 (0.675) | -1.43 (0.554)
  Week 12 after second injection in OL | -1.19 (0.732) | -1.21 (0.750)
  Week 4 after third injection in OL | -1.48 (0.750) | -1.43 (0.764)
  Week 8 after third injection in OL | -1.41 (0.694) | -1.43 (0.556)
  Week 12 after third injection in OL | -1.44 (0.751) | -1.34 (0.578)

9. Secondary Outcome: Mean Change From Baseline (at the Start of the Double-blind Phase) in the Physician's Rating Score (PRS) at 4, 8, and 12 Weeks After Each Injection in the Open-label Phase
Description: The investigator assessed the PRS of gait pattern consisting of 3 parameters. Affected limb was scored on a scale of -1 (worst) to 9 (best) based on 3 parameters (initial foot contact, foot contact at midstance, gait assistive devices) at each time point from baseline (at the start of the double-blind phase) to Week 48.
Time Frame: Baseline; Weeks 4, 8, and 12 after each injection (up to Week 48; injections given from Week 12 to Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | DB BTX + OL BTX | DB Placebo + OL BTX
Number analyzed (Participants) | 50 | 57
Points on a scale
  Week 4 after first injection in OL | 1.10 (1.433) | 1.35 (1.601)
  Week 8 after first injection in OL | 1.17 (1.494) | 1.46 (1.668)
  Week 12 after first injection in OL | 0.91 (1.501) | 1.15 (1.638)
  Week 4 after second injection in OL | 1.30 (1.389) | 1.48 (1.722)
  Week 8 after second injection in OL | 1.33 (1.569) | 1.47 (1.700)
  Week 12 after second injection in OL | 1.40 (1.449) | 1.29 (1.842)
  Week 4 after third injection in OL | 1.28 (1.461) | 1.04 (1.551)
  Week 8 after third injection in OL | 1.33 (1.494) | 1.15 (1.433)
  Week 12 after third injection in OL | 1.22 (1.121) | 0.96 (1.344)

10. Secondary Outcome: Mean Change From Baseline (at the Start of the Double-blind Phase) in the Time (Seconds) to Walk 10 Meters at 4, 8, and 12 Weeks After Each Injection in the Open-label Phase
Description: The time (seconds) required to walk 10 meters was measured at each time point from baseline (at the start of the double-blind phase) to Week 48.
Time Frame: Baseline; Weeks 4, 8, and 12 after each injection (up to Week 48; injections given from Week 12 to Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | DB BTX + OL BTX | DB Placebo + OL BTX
Number analyzed (Participants) | 50 | 57
seconds
  Week 4 after first injection in OL | -11.21 (25.670) | -12.09 (27.148)
  Week 8 after first injection in OL | -11.14 (27.453) | -8.05 (22.735)
  Week 12 after first injection in OL | -10.50 (27.726) | -9.29 (21.851)
  Week 4 after second injection in OL | -13.49 (29.674) | -13.05 (31.241)
  Week 8 after second injection in OL | -8.05 (45.061) | -7.65 (22.715)
  Week 12 after second injection in OL | -16.31 (32.613) | -13.40 (29.508)
  Week 4 after third injection in OL | -20.09 (42.452) | -13.42 (33.205)
  Week 8 after third injection in OL | -15.91 (43.589) | -12.10 (28.240)
  Week 12 after third injection in OL | -16.37 (51.482) | -13.84 (29.241)

11. Secondary Outcome: Mean Change From Baseline (at the Start of the Double-blind Phase) in the Clinical Global Impression (CGI) Score of Functional Disability Assessed by the Investigator at 4, 8, and 12 Weeks After Each Injection in the Open-label Phase
Description: The CGI of functional disability was assessed at each visit using the 11-point Numeric Rating Scale (NRS) (-5=Worst Possible to 5=Best Possible) at each time point from baseline (at the start of the double-blind phase) to Week 48.
Time Frame: Baseline; Weeks 4, 8, and 12 after each injection (up to Week 48; injections given from Week 12 to Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | DB BTX + OL BTX | DB Placebo + OL BTX
Number analyzed (Participants) | 50 | 57
Points on a scale
  Week 4 after first injection in OL | 1.43 (1.443) | 1.43 (1.463)
  Week 8 after first injection in OL | 1.40 (1.393) | 1.54 (1.513)
  Week 12 after first injection in OL | 1.11 (1.387) | 1.21 (1.589)
  Week 4 after second injection in OL | 1.93 (1.639) | 2.02 (1.550)
  Week 8 after second injection in OL | 1.70 (1.670) | 1.89 (1.676)
  Week 12 after second injection in OL | 1.55 (1.611) | 1.52 (1.683)
  Week 4 after third injection in OL | 2.07 (1.387) | 1.59 (1.476)
  Week 8 after third injection in OL | 2.04 (1.224) | 1.82 (1.389)
  Week 12 after third injection in OL | 2.00 (1.177) | 1.68 (1.416)

12. Secondary Outcome: Mean Change From Baseline (at the Start of the Double-blind Phase) in the Clinical Global Impression (CGI) Score of Functional Disability Assessed by the Participant at 4, 8, and 12 Weeks After Each Injection in the Open-label Phase
Description: as for outcome 11
Time Frame: Baseline; Weeks 4, 8, and 12 after each injection (up to Week 48; injections given from Week 12 to Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | DB BTX + OL BTX | DB Placebo + OL BTX
Number analyzed (Participants) | 50 | 57
Points on a scale
  Week 4 after first injection in OL | 0.92 (1.891) | 1.00 (2.149)
  Week 8 after first injection in OL | 0.98 (2.080) | 1.04 (2.215)
  Week 12 after first injection in OL | 0.66 (1.536) | 1.19 (2.349)
  Week 4 after second injection in OL | 1.26 (2.205) | 1.75 (1.973)
  Week 8 after second injection in OL | 1.37 (2.226) | 1.67 (2.119)
  Week 12 after second injection in OL | 1.19 (2.222) | 1.57 (2.029)
  Week 4 after third injection in OL | 1.62 (2.305) | 1.66 (1.396)
  Week 8 after third injection in OL | 1.56 (2.532) | 1.86 (1.715)
  Week 12 after third injection in OL | 1.33 (2.557) | 1.86 (2.013)

13. Secondary Outcome: Mean Change From Baseline (at the Start of the DB Phase) in the Clinical Global Impression (CGI) Score of Functional Disability Assessed by the Physiotherapist/Occupational Therapist at 4, 8, and 12 Weeks After Each Injection in the Open-label Phase
Description: as for outcome 11
Time Frame: Baseline; Weeks 4, 8, and 12 after each injection (up to Week 48; injections given from Week 12 to Week 36)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | DB BTX + OL BTX | DB Placebo + OL BTX
Number analyzed (Participants) | 50 | 57
Points on a scale
  Week 4 after first injection in OL | 1.14 (1.708) | 1.54 (1.878)
  Week 8 after first injection in OL | 1.40 (1.814) | 1.54 (1.768)
  Week 12 after first injection in OL | 1.28 (1.919) | 1.46 (1.702)
  Week 4 after second injection in OL | 1.49 (1.882) | 2.00 (1.798)
  Week 8 after second injection in OL | 1.42 (1.880) | 1.76 (1.888)
  Week 12 after second injection in OL | 1.57 (1.965) | 1.83 (1.992)
  Week 4 after third injection in OL | 1.38 (1.840) | 1.62 (2.145)
  Week 8 after third injection in OL | 1.30 (1.918) | 1.86 (2.155)
  Week 12 after third injection in OL | 1.59 (2.438) | 1.50 (2.219)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were classified by onset time because the study consists of the double-blind (DB) and open-label (OL) phases.
Description: AEs in the double-blind (DB) phase (Arms 1-2), AEs occurring after the start (injection) of the DB phase (Week 0), but before the first injection day in the open-label (OL) phase; AEs in the OL phase (Arms 3-4), AEs occurring after the first injection day in the OL phase. SAEs and AEs were analyzed in the Full Analysis Set.
Arm/Group | BTX 300U | Placebo | DB BTX + OL BTX | DB Placebo + OL BTX
Serious Adverse Events (participants affected / at risk) | 5/58 | 1/62 | 3/50 | 8/57
Other Adverse Events (participants affected / at risk) | 16/58 | 16/62 | 23/50 | 16/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BTX 300U (N=58) | Placebo (N=62) | DB BTX + OL BTX (N=50) | DB Placebo + OL BTX (N=57)
Angina pectoris (Cardiac disorders) | 2 | 0 | 0 | 0
Gastric ulcer hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Mania (Psychiatric disorders) | 0 | 0 | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BTX 300U (N=58) | Placebo (N=62) | DB BTX + OL BTX (N=50) | DB Placebo + OL BTX (N=57)
Nasopharyngitis (Infections and infestations) | 8 | 12 | 15 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 0
Injection site pain (General disorders) | 3 | 1 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 0 | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 5 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 1 | 3 | 3
Pyrexia (General disorders) | 0 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.